CLINICAL TRIAL: NCT06510465
Title: Neoadjuvant Therapy With Weekly Utidelone Combined With Cisplatin for Patients With Breast Cancer (NeoURANIA): A Multi-center, Prospective Study
Brief Title: Neoadjuvant Therapy With Weekly Utidelone Combined With Cisplatin for Patients With Breast Cancer (NeoURANIA)
Acronym: NeoURANIA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHPD009
Record Dates: First submitted 2024-05-23; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; utidelone; cisplatin; neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Cisplatin; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HER2 negative breast cancer cohort (Experimental): Human Epidermal Growth Factor Receptor 2 (HER2 ) negative breast cancer utidelone and cisplatin
  Interventions: Drug: utidelone; Drug: Cisplatin
- HER2 positive breast cancer cohort (Experimental): Human Epidermal Growth Factor Receptor 2 (HER2 ) positive breast cancer utidelone，cisplatin，tratuzumab and pertuzumab (both Intravenous preparations or subcutaneous preparations can be used)
  Interventions: Drug: utidelone; Drug: Cisplatin; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: utidelone — utidelone 50mg／m2，ivgtt，d1，8，15，22, q28d, up to 4 cycle；
  Other Names: UTD1
Drug: Cisplatin — cisplatin25mg/m2，ivgtt，d1，8，15；q28d, up to 4 cycle.
  Other Names: DDP
Drug: Trastuzumab — Trastuzumab 8mg/kg, ivgtt, d1, then 6mg/kg, q21d or Trastuzumab 4mg/kg, ivgtt, d1, then 2mg/kg, q7d or Trastuzumab Injection（Subcutaneous Injection）600mg，subcutaneous Injection，d1，q21d
  Arms: HER2 positive breast cancer cohort
Drug: Pertuzumab — Pertuzumab 840mg, ivgtt, d1, then 420mg, q21d or Pertuzumab/trastuzumab/hyaluronidase
  Arms: HER2 positive breast cancer cohort

SUMMARY:
This study is a prospective, multi-center, single-arm, two-cohort, exploratory study, aiming to explore the effectiveness and safety of neoadjuvant treatment with weekly utidelone combined with cisplatin in breast cancer patients.

DETAILED DESCRIPTION:
Explore the effectiveness and safety of neoadjuvant treatment with weekly utidelone combined with cisplatin in high risk early, locally advanced and Inflammatory breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Primary invasive breast cancer confirmed by pathology; Before neoadjuvant therapy, the primary breast lesion was larger than 2cm(cT2-T4a-d, according to the anatomical staging of AJCC 8th edition), or the clinical images of lymph nodes considered metastasis or pathologically confirmed metastasis (CN+); or patients whose primary breast lesions are more than 1cm and less than 2cm, and whose lymph nodes have not metastasized (cT1cN0) must meet one of the following conditions: hormone receptor negative, HER2 positive, or ki67 greater than 20%. If bilateral breast cancer is found at the same time, it can be admitted to the group, but it is necessary to determine which side of the lesion is to be evaluated before taking the drug;
3. According to the RECIST version 1.1 standard (see Annex I), there is at least one measurable lesion before neoadjuvant therapy;
4. The score of ECOG is 0 or 1;
5. During neoadjuvant therapy, ovarian function suppression can be given at the same time;
6. The hematological examination and blood biochemical examination should meet the following requirements: white blood cell count (WBC)≥3.0×109/L, neutrophil count (ANC)≥1.5×109/L and platelet count (PLT) ≥ 75× 109/L; Hemoglobin (HB) ≥ 80g/L; Total bilirubin (TBIL)≤1.5× upper limit of normal value (ULN), AST(sGOT), ALT(sGPT)≤2×ULN and creatinine (Cr) ≤ 1.5× ULN;
7. creatinine clearance rate ≥50mL/min(Cockcroft-Gault formula);
8. Subjects voluntarily joined the study, signed the informed consent form, and had good compliance and cooperated with the follow-up.

Exclusion Criteria:

1. Patients during pregnancy and lactation, patients with fertility and positive baseline pregnancy test, or women of childbearing age who are unwilling to take effective contraceptive measures during the whole trial period;
2. There is distant metastasis of breast cancer confirmed by imaging or pathology before enrollment;
3. There is evidence of sensory or motor nerve diseases;
4. Severe cardiopulmonary insufficiency, severe hepatic and renal insufficiency, severe concomitant disease or active infection, including known HIV infection;
5. allergic to the research drug or its auxiliary materials;
6. Arterial/venous thrombotic events, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, occurred within 6 months before the start of the study;
7. Previous history of other malignant tumors, except the cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and the second primary malignant tumor with high 5-year recurrence-free survival rate determined by researchers;
8. According to the researcher's judgment, there are accompanying diseases (including but not limited to uncontrollable hypertension, severe diabetes, active infection, thyroid disease, etc.) that seriously endanger the patient's safety or affect the patient's completion of the study, and any other circumstances that the researcher judges that the patient is not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
pCR | through surgery completion, an average of 16 weeks
  ypT0/is ypN0

SECONDARY OUTCOMES:
breast pCR | through surgery completion, an average of 16 weeks
  ypT0/is
RCB 0/I rate | through surgery completion, an average of 16 weeks
  ratio of patients who achieved RCB 0 or RCB I
RCB class | through surgery completion, an average of 16 weeks
  RCB 0, RCB I, RCB II, RCB III
Rate of lymph node negative | through surgery completion, an average of 16 weeks
  ratio of patients who achieved lymph node negative
ORR by physical examination | After completing neoadjuvant therapy before surgery, an average of 16 weeks
  ratio of patients who achieved complete response or partial response by physical examination
ORR by MRI | After completing neoadjuvant therapy before surgery, an average of 16 weeks
  ratio of patients who achieved complete response or partial response by MRI
CBR by physical examination | After completing neoadjuvant therapy before surgery, an average of 16 weeks
  ratio of patients who achieved complete response or partial response or stable disease by physical examination
CBR by MRI | After completing neoadjuvant therapy before surgery, an average of 16 weeks
  ratio of patients who achieved complete response or partial response or stable disease by MRI
iDFS | 2year,3year,5year,8year,10year
  It is defined as the time from first dose of study intervention administration to the first occurrence of ipsilateral invasive cancer recurrence, contralateral invasive breast cancer, local and/or regional invasive cancer recurrence, distant metastasis or death from any cause.
EFS | 2year,3year,5year,8year,10year
  It is defined as the time from first dose of study intervention administration to the first occurrence of local and/or regional recurrence, contralateral breast cancer, distant metastasis or death from any cause.
DDFS | 2year,3year,5year,8year,10year
  It is defined as the time from first dose of study intervention administration to the first distant metastasis or death from any cause.
OS | 2year,3year,5year,8year,10year
  It is defined as the time from first dose of study intervention administration to death from any cause.
Quality of Life | Through study completion，an average of 1 year
  EORTC-QLQ-C30
Quality of Life | Through study completion，an average of 1 year
  EORTC-QLQ-BR23
Safety | Through study completion，an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Combine with weekly paclitaxel with cispltin in HER2-negative and HER2-positive patients | After completing neoadjuvant therapy before surgery, an average of 16 weeks
  Combine with weekly paclitaxel with cispltin in HER2-negative and HER2-positive patients

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No